CLINICAL TRIAL: NCT01411891
Title: Prospective Randomized Control Trial of Post-Operative Colonization Rates of Femoral Nerve Catheters With the Use of Chlorhexidine-Impregnated Patch
Brief Title: Post-Operative Colonization Rates of Femoral Nerve Catheters Treated With Chlorhexidine-Impregnated Patch
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-0444
Record Dates: First submitted 2011-05-17; First posted 2011-08-08 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Catheter Infections; Spinal Catheter (Epidural) (Subdural); Complications, Infection or Inflammation
Keywords: Arthroplasty; Infection Control
MeSH Terms: conditions — Infections; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients assigned to this study group will not have a chlorhexidine impregnated patch placed at the femoral nerve catheter insertion site.
- Chlorhexidine impregnated patch. (Experimental): Patients assigned to this study group will have a chlorhexidine impregnated patch placed at the femoral nerve catheter insertion site.
  Interventions: Device: Chlorhexidine impregnated patch (Biopatch)

INTERVENTIONS:
Device: Chlorhexidine impregnated patch (Biopatch) — Patients assigned to the intervention group will have a chlorhexidine impregnated patch placed at the femoral nerve catheter insertion site.
  Other Names: Biopatch
  Arms: Chlorhexidine impregnated patch.

SUMMARY:
Joint replacement is becoming an increasingly common procedure. In 2005, 534,000 total knee arthroplasties (TKA) were performed in the United States which is at a rate of 18.1 per 10,000 individuals, and the demand for primary TKA is projected to grow by 673% by 2030. Effective post-operative analgesia is an important component with regards to patient satisfaction and hospital stay. Regional anesthesia has been shown to decrease duration of surgery, need for transfusion, post-operative nausea and vomiting, and the incidence of thromboembolic disease in patients undergoing total knee or total hip replacement when compared with general anesthesia. Post-operatively, regional anesthesia has been shown to reduce pain scores and/or morphine consumption as well as opioid-related adverse effects.

Epidural catheter or spinal anesthesia has become the standard of care at the University of Wisconsin-Madison for intraoperative management of TKA patients. General anesthesia is still occasionally used for patients that would strongly prefer a general anesthetic, those that are taking anticoagulation medications or with a coagulopathy, those with previous back surgery, and those with certain neurologic conditions such as multiple sclerosis or spina bifida. Comparison studies between lumbar epidural analgesia and femoral nerve catheters (FNC) for postoperative analgesia following TKA show no significant difference in pain scores, morphine consumption, or post-operative nausea and vomiting. However, epidural analgesia has been associated with higher incidence of hypotension and urinary retention. FNC's placed for postoperative pain allow patients to ambulate more effectively as there should not be much of a lower extremity motor block. Patients with a FNC for postoperative analgesia also do not require a urinary catheter which eliminates a common source of infection in postoperative patients. FNCs have also demonstrated improved rehabilitation times and decreased hospital stays which has led to an increased insertion rate of FNCs for postoperative analgesia following TKA at the University of Wisconsin.

Pyarthrosis is a fairly common complication occurring at a rate of 2% following primary and 5.6% following revision TKA. Infection can be a devastating complication following implantation of joint hardware often leading to extended hospitalization/rehabilitation stays and return trips to the operating room. The average billed charges for all types of revision TKA procedures was $49,360 with average length of stay of 5.1 days. Indwelling lines are a known infection risk and indwelling lines in the femoral region are known to be associated with a high incidence of catheter colonization. At 48 hours, Cuvillon et. al. found that 57% of FNCs placed without the use of a chlorhexidine impregnated patch had positive bacterial colonization. They also described three cases of transient bacteremia secondary to FNCs in the 208 catheters that they analyzed.

Chlorhexidine impregnated patches also known as "biopatches" have been shown to reduce the incidence of bacterial colonization and infection of various indwelling lines including epidurals and central venous catheters. Currently no standard of care exists that requires the use of biopatches for FNCs. The investigators propose studying the use of the biopatch to reduce the incidence of bacterial colonization of femoral nerve catheters.

The investigators will study the efficacy of the biopatch at decreasing the rate of bacterial colonization of FNCs in TKA patients. The FNCs will be inserted in the standard fashion and removed at the end of therapy. Typically the FNC infusion will continue until the morning of post-operation day (POD) #1 or 2. The process for FNC insertion first involves sterile prep and drape of the femoral region. Full sterile technique will be utilized including gown, gloves, and mask. Ultrasound guidance is then commonly utilized to identify the femoral nerve. Following patient sedation and skin infiltration with local anesthetic, a tuohy needle is inserted adjacent to the femoral nerve. A catheter is then threaded through the needle in close proximity to the femoral nerve. Patients will be randomized to either no chlorhexidine impregnated patch or to a chlorhexidine impregnated patch that will be located at the catheter exit site. On the morning of POD 1 or 2, the FNC infusion will be discontinued. Typically, Twenty-four to forty-eight hours after catheter insertion, it will be removed in a sterile fashion and the skin surrounding the catheter exit site will be swabbed and the distal catheter tip will be sent for culture to determine bacterial colonization. In addition, the investigators will interview patients and review clinical data to determine signs of infection and/or catheter tip colonization rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-85 undergoing elective knee arthroplasty who elect to have a femoral nerve block catheter placed for postoperative analgesia.

Exclusion Criteria:

* Allergy to local anesthetics,
* local or generalized infection or inflammation,
* current antibiotic therapy,
* immunocompromised patients,
* a history of chronic steroid use,
* neurological deficits,
* pregnancy,
* prisoners,
* refusal to participate,
* primary language other than English,
* and patients currently participating in a study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristopher M Schroeder, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Result] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Result] Hu S, Zhang ZY, Hua YQ, Li J, Cai ZD. A comparison of regional and general anaesthesia for total replacement of the hip or knee: a meta-analysis. J Bone Joint Surg Br. 2009 Jul;91(7):935-42. doi: 10.1302/0301-620X.91B7.21538. PMID 19567860
- [Result] Macfarlane AJ, Prasad GA, Chan VW, Brull R. Does regional anesthesia improve outcome after total knee arthroplasty? Clin Orthop Relat Res. 2009 Sep;467(9):2379-402. doi: 10.1007/s11999-008-0666-9. Epub 2009 Jan 7. PMID 19130163
- [Result] Fowler SJ, Symons J, Sabato S, Myles PS. Epidural analgesia compared with peripheral nerve blockade after major knee surgery: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2008 Feb;100(2):154-64. doi: 10.1093/bja/aem373. PMID 18211990
- [Result] Konig DP, Schierholz JM, Munnich U, Rutt J. Treatment of staphylococcal implant infection with rifampicin-ciprofloxacin in stable implants. Arch Orthop Trauma Surg. 2001 May;121(5):297-9. doi: 10.1007/s004020000242. PMID 11409564
- [Result] Bozic KJ, Kurtz SM, Lau E, Ong K, Chiu V, Vail TP, Rubash HE, Berry DJ. The epidemiology of revision total knee arthroplasty in the United States. Clin Orthop Relat Res. 2010 Jan;468(1):45-51. doi: 10.1007/s11999-009-0945-0. Epub 2009 Jun 25. PMID 19554385
- [Result] Cuvillon P, Ripart J, Lalourcey L, Veyrat E, L'Hermite J, Boisson C, Thouabtia E, Eledjam JJ. The continuous femoral nerve block catheter for postoperative analgesia: bacterial colonization, infectious rate and adverse effects. Anesth Analg. 2001 Oct;93(4):1045-9. doi: 10.1097/00000539-200110000-00050. PMID 11574381
- [Result] Compere V, Legrand JF, Guitard PG, Azougagh K, Baert O, Ouennich A, Fourdrinier V, Frebourg N, Dureuil B. Bacterial colonization after tunneling in 402 perineural catheters: a prospective study. Anesth Analg. 2009 Apr;108(4):1326-30. doi: 10.1213/ane.0b013e31819673aa. PMID 19299807
- [Result] Ho KM, Litton E. Use of chlorhexidine-impregnated dressing to prevent vascular and epidural catheter colonization and infection: a meta-analysis. J Antimicrob Chemother. 2006 Aug;58(2):281-7. doi: 10.1093/jac/dkl234. Epub 2006 Jun 6. PMID 16757502
- [Result] Mann TJ, Orlikowski CE, Gurrin LC, Keil AD. The effect of the biopatch, a chlorhexidine impregnated dressing, on bacterial colonization of epidural catheter exit sites. Anaesth Intensive Care. 2001 Dec;29(6):600-3. doi: 10.1177/0310057X0102900606. PMID 11771602
- [Result] Morin AM, Kerwat KM, Klotz M, Niestolik R, Ruf VE, Wulf H, Zimmermann S, Eberhart LH. Risk factors for bacterial catheter colonization in regional anaesthesia. BMC Anesthesiol. 2005 Mar 17;5(1):1. doi: 10.1186/1471-2253-5-1. PMID 15774007
- [Result] Shapiro JM, Bond EL, Garman JK. Use of a chlorhexidine dressing to reduce microbial colonization of epidural catheters. Anesthesiology. 1990 Oct;73(4):625-31. doi: 10.1097/00000542-199010000-00007. PMID 2121070
- [Result] Yuan HB, Zuo Z, Yu KW, Lin WM, Lee HC, Chan KH. Bacterial colonization of epidural catheters used for short-term postoperative analgesia: microbiological examination and risk factor analysis. Anesthesiology. 2008 Jan;108(1):130-7. doi: 10.1097/01.anes.0000296066.79547.f3. PMID 18156891
- [Derived] Schroeder KM, Jacobs RA, Guite C, Gassner K, Anderson B, Donnelly MJ. Use of a chlorhexidine-impregnated patch does not decrease the incidence of bacterial colonization of femoral nerve catheters: a randomized trial. Can J Anaesth. 2012 Oct;59(10):950-7. doi: 10.1007/s12630-012-9768-7. Epub 2012 Aug 2. PMID 22855310

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Chlorhexidine Impregnated Patch.
Started | 50 | 50
Completed | 47 | 48
Not Completed | 3 | 2
Not completed — Catheter dislodgement or loss to follow- | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Chlorhexidine Impregnated Patch. | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 37 | 63
  >=65 years | 21 | 11 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.6) | 61.2 (8.6) | 63 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 28 | 24 | 52
Region of Enrollment [Number; unit: participants]
  United States | 47 | 48 | 95

OUTCOME MEASURES:

1. Primary Outcome: Catheter Tip Colonization
Description: Three cm of the for research purposes only, a 3 cm distal portion will be cut using sterile scissors into a sterile container, and sent to the lab for culture in a sterile container. The catheter segments will be rolled onto blood agar plates at 35°C under aerobic and anaerobic conditions. Number of colonies will be counted at 1 week. The peripheral nerve catheter tip will be considered colonized if the culture yields 15 or greater colony forming units.
Time Frame: 24-48 hours after placement of femoral nerve catheter.
Population: Patients presenting for elective TKA.
Measure: Number; unit: participants
Arm/Group | Control | Chlorhexidine Impregnated Patch.
Number analyzed (Participants) | 47 | 48
participants | 2 | 3
Statistical Analysis 1: Comparison: Control vs Chlorhexidine Impregnated Patch; Test type: Superiority; Risk Ratio (RR) = 1.5, 95% CI 2-sided [0.3 to 8.4]

2. Secondary Outcome: Catheter Insertion Site Colonization.
Description: Skin at the FNC insertion site will be swabbed with a sterile cotton tip applicator moistened with sterile normal saline. The swab will be placed in a sterile container. The swab will be inoculated onto a blood agar plate/eosin-methylene blue plate/chocolate agar plate and incubated for 3 days aerobically, then inoculated onto an anaerobic brucella-agar plate and incubated for 7 days anaerobically. Bacterial growth found in the first quadrant of the inoculated plate will be defined as low grade, in the second and/or third will be moderate, and in the fourth quadrant will be heavy.
Time Frame: 24-48 hours.
Measure: Number; unit: participants
Arm/Group | Control | Chlorhexidine Impregnated Patch.
Number analyzed (Participants) | 47 | 48
participants | 14 | 12
Statistical Analysis 1: Comparison: Control vs Chlorhexidine Impregnated Patch; Test type: Superiority; p = 0.65, Regression, Logistic; Risk Ratio (RR) = 0.8, 95% CI 2-sided [0.4 to 1.6]

ADVERSE EVENTS:
Arm/Group | Control | Chlorhexidine Impregnated Patch.
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 0/47 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes